CLINICAL TRIAL: NCT05924971
Title: Acetylsalicylic Acid for Postpartum Preeclampsia: A Pilot Randomized Trial
Brief Title: Aspirin for Postpartum Patients With Preeclampsia
Acronym: ASAPP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Collaborators: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Megan Oakes, MD MSCI, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 371-23
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia Postpartum
Keywords: Preeclampsia; Postpartum; Aspirin; sFlt-1
MeSH Terms: conditions — Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Patients with preeclampsia will be randomized after delivery to receive either standard blood pressure control plus aspirin 81 mg or standard blood pressure control alone.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor will be blinded to study arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard blood pressure control plus aspirin 81 mg (Experimental): Standardized postpartum blood pressure control Aspirin 81 mg by mouth x 1 week post-delivery
  Interventions: Drug: Aspirin 81Mg Ec Tab
- Standard blood pressure control (No Intervention): Standardized postpartum blood pressure control

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab — Aspirin 81 mg 1 tablet by mouth. Participants randomized to receive aspirin in addition to standard blood pressure management will receive the study medication nightly at 20:00, with first dose initiated within 24 hours of delivery.
  Arms: Standard blood pressure control plus aspirin 81 mg

SUMMARY:
The purpose of this research study is to evaluate the effect of low-dose aspirin on recovery from severe preeclampsia (a high blood pressure disorder of pregnancy) among women who have given birth. We hypothesize that taking aspirin for the first week after giving birth will enhance recovery from preeclampsia by decreasing the levels of a protein called soluble fms-like tyrosine kinase (sFlt-1), which is thought to be a main contributor to the development of preeclampsia, and speeding up return to a normal blood pressure.

DETAILED DESCRIPTION:
Preeclampsia is a condition of the antenatal and postpartum periods, which manifests as new-onset hypertension and end-organ damage. Globally, preeclampsia is estimated to affect up to 9% of all pregnancies, though as many as two-thirds of patients who receive this diagnosis will remain hypertensive beyond the time of their postpartum hospital discharge. Because of this, postpartum preeclampsia is the leading cause of postpartum hospital readmission in the United States. Anti-hypertensive medications and magnesium sulfate are temporizing therapies aimed at preventing the immediate sequelae of preeclampsia such as seizures, stroke, and end-organ damage. However, there are no therapies directly targeting the pathophysiology underlying postpartum preeclampsia, which poses difficulties in promoting blood pressure recovery to a normotensive state.

Preeclampsia is considered a disorder of abnormal placentation, leading to the release of abnormal pro-angiogenic, anti-angiogenic, and vasoactive molecules. Specifically, excess elevations in anti-angiogenic proteins like soluble fms-like tyrosine kinase 1 (sFlt-1) relative to pro-angiogenic proteins like placental growth factor (PlGF) are thought to cause vasospasm and, in turn, hypertension. As such, it seems plausible that persistent postpartum sFlt-1 elevation is implicated in the pathophysiology of postpartum preeclampsia.

At low doses, acetylsalicylic acid, or aspirin, has been proven to target the aforementioned angiogenic imbalance by decreasing serum sFlt-1 levels. While aspirin is widely used during pregnancy to mitigate the risk of preeclampsia, the utility of aspirin in the postpartum period to target these pathways and promote BP recovery to a normotensive state is unknown. The central hypothesis of this trial is that use of aspirin in the first week postpartum will enhance recovery from preeclampsia by improving blood pressure recovery via decreased levels of sFlt-1.

ELIGIBILITY:
Inclusion Criteria:

* Preeclampsia with severe features diagnosed during delivery admission, as defined by ACOG criteria.
* Pre- and postnatal care provided by the Long Beach Memorial Ob/Gyn resident or Maternal-Fetal Medicine clinic.

Exclusion Criteria:

* Patient age <18 years old
* Non-English or Non-Spanish speaking
* Chronic hypertension diagnosed before 20 weeks' gestation
* Known allergy, prior adverse reaction, or any medical condition in which aspirin is contraindicated (nasal polyps, gastric or duodenal ulcers, history of gastrointestinal bleeding, severe hepatic dysfunction)
* Aspirin prescribed postpartum for any other medical condition
* Bleeding disorder
* Breastfeeding an infant with thrombocytopenia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in sFlt-1 | 1 week postpartum
  This outcome will determine the absolute change in sFlt-1, an anti-angiogenic protein implicated in the pathophysiology of preeclampsia.

SECONDARY OUTCOMES:
Normotension (ACOG) | 1 week postpartum
  This outcome will measure the proportion of patients who achieve a blood pressure of <140/90, as defined by ACOG, without any further elevated values.
Normotension (JNC) | 1 week postpartum
  This outcome will measure the proportion of patients who achieve a blood pressure of <130/80, as defined by JNC, without any further elevated values.
Time to normotension | 6 weeks postpartum
  This outcome will assess the length of time in days to normotension after randomization. Normotension will be defined by both ACOG and JNC criteria.
Anti-hypertensive therapy | 6 weeks postpartum
  This outcome will assess if additional or increased doses of anti-hypertensive therapies are needed following randomization.
Readmission | 6 weeks postpartum
  This outcome will assess if a study participant is readmitted for blood pressure or preeclampsia related reasons following randomization.
Adherence | 1 week postpartum
  This outcome will assess for adherence to aspirin therapy in those randomized to the aspirin arm. This is defined as greater than 90% consumption of the prescribed doses.
Enrollment feasibility | 1 week postpartum
  This outcome will assess feasibility for future studies, defined as both the number of patients randomized by the number of patients eligible and the number of patients who completed the study protocol divided by the number of patients randomized.
Postpartum hemorrhage | 6 weeks postpartum
  This safety outcome is defined as a postpartum hemorrhage of greater than 1 liter following randomization.
Postpartum bleeding requiring intervention | 6 weeks postpartum
  This safety outcome is defined as postpartum bleeding requiring intervention (uterotonic administration, intrauterine balloon placement, dilation and curettage, or uterine artery embolization) following randomization.
Unplanned postpartum evaluation for bleeding | 6 weeks postpartum
  This safety outcome is defined as the need for urgent evaluation for bleeding in the clinic/office, obstetrical triage unit, or emergency room for vaginal bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Megan C Oakes, MD MSCI, Principal Investigator — Miller Children's and Women's Hospital, Long Beach/ MemorialCare Medical Center
Locations (1):
- Miller Children's and Women's Hospital, Long Beach/MemorialCare Long Beach, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 202: Gestational Hypertension and Preeclampsia. Obstet Gynecol. 2019 Jan;133(1):1. doi: 10.1097/AOG.0000000000003018. PMID 30575675
- [Background] Ditisheim A, Wuerzner G, Ponte B, Vial Y, Irion O, Burnier M, Boulvain M, Pechere-Bertschi A. Prevalence of Hypertensive Phenotypes After Preeclampsia: A Prospective Cohort Study. Hypertension. 2018 Jan;71(1):103-109. doi: 10.1161/HYPERTENSIONAHA.117.09799. Epub 2017 Nov 13. PMID 29133363
- [Background] Mogos MF, Salemi JL, Spooner KK, McFarlin BL, Salihu HH. Hypertensive disorders of pregnancy and postpartum readmission in the United States: national surveillance of the revolving door. J Hypertens. 2018 Mar;36(3):608-618. doi: 10.1097/HJH.0000000000001594. PMID 29045342
- [Background] Agrawal S, Cerdeira AS, Redman C, Vatish M. Meta-Analysis and Systematic Review to Assess the Role of Soluble FMS-Like Tyrosine Kinase-1 and Placenta Growth Factor Ratio in Prediction of Preeclampsia: The SaPPPhirE Study. Hypertension. 2018 Feb;71(2):306-316. doi: 10.1161/HYPERTENSIONAHA.117.10182. Epub 2017 Dec 11. PMID 29229743
- [Background] Su MT, Wang CY, Tsai PY, Chen TY, Tsai HL, Kuo PL. Aspirin enhances trophoblast invasion and represses soluble fms-like tyrosine kinase 1 production: a putative mechanism for preventing preeclampsia. J Hypertens. 2019 Dec;37(12):2461-2469. doi: 10.1097/HJH.0000000000002185. PMID 31335509
- [Background] Lin L, Li G, Zhang W, Wang YL, Yang H. Low-dose aspirin reduces hypoxia-induced sFlt1 release via the JNK/AP-1 pathway in human trophoblast and endothelial cells. J Cell Physiol. 2019 Aug;234(10):18928-18941. doi: 10.1002/jcp.28533. Epub 2019 Apr 19. PMID 31004367
- [Background] Neuman RI, Figaroa AMJ, Nieboer D, Saleh L, Verdonk K, Danser AHJ, Duvekot HJJ, van den Meiracker AH, Roeters van Lennep J, Visser W. Angiogenic markers during preeclampsia: Are they associated with hypertension 1 year postpartum? Pregnancy Hypertens. 2021 Mar;23:116-122. doi: 10.1016/j.preghy.2020.11.011. Epub 2020 Dec 3. PMID 33321329
- [Background] Whelton PK, Carey RM, Aronow WS, Casey DE Jr, Collins KJ, Dennison Himmelfarb C, DePalma SM, Gidding S, Jamerson KA, Jones DW, MacLaughlin EJ, Muntner P, Ovbiagele B, Smith SC Jr, Spencer CC, Stafford RS, Taler SJ, Thomas RJ, Williams KA Sr, Williamson JD, Wright JT Jr. 2017 ACC/AHA/AAPA/ABC/ACPM/AGS/APhA/ASH/ASPC/NMA/PCNA Guideline for the Prevention, Detection, Evaluation, and Management of High Blood Pressure in Adults: Executive Summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Hypertension. 2018 Jun;71(6):1269-1324. doi: 10.1161/HYP.0000000000000066. Epub 2017 Nov 13. No abstract available. PMID 29133354